CLINICAL TRIAL: NCT03175315
Title: Evaluation of a Newly Developed Psychoeducational Treatment and Education Program for People With Type 1 and Type 2 Diabetes on an Intensified Insulin Therapy Who Use Flash Glucose Monitoring
Brief Title: Evaluation of a Treatment and Education Program for Diabetic Patients Who Use Flash Glucose Monitoring
Acronym: FLASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norbert Hermanns (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor-Investigator, Norbert Hermanns, CEO, Forschungsinstitut der Diabetes Akademie Mergentheim
Organization: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH052017
Record Dates: First submitted 2017-05-02; First posted 2017-06-05 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus
Keywords: psychoeducation; treatment and education programme; self-management; diabetes education; flash glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLASH (Experimental): Intervention: Conduct of the newly developed treatment and education program for patients with diabetes who use flash glucose monitoring (FLASH).
  FLASH consists of 4 lessons focusing on empowering patients to autonomously use flash glucose monitoring (FGM) in their daily routine. Patients learn to effectively interpret the different information provided by FGM in order to improve not only glycemic control but also to improve the implementation of insulin therapy in daily life. Psychological and motivational aspects of living with diabetes and handling of the FGM are addressed as well.
  Interventions: Behavioral: Treatment and education program for patients with diabetes who use flash glucose monitoring (FLASH)
- Waiting List (No Intervention): Diabetic patients using FGM receive treatment as usual until the last measurement point. After completion of the study, they are offered participation in the FLASH program.

INTERVENTIONS:
Behavioral: Treatment and education program for patients with diabetes who use flash glucose monitoring (FLASH) — Treatment and education program based on the self-management theory of behavioral medicine. The program is delivered by certified and specially trained diabetes educators.
  Arms: FLASH

SUMMARY:
This study is a randomized, controlled, prospective trial with a 6-month follow- up. A newly developed psychoeducational treatment and education programme for diabetic patients on an insulin therapy who use flash glucose monitoring (FGM) will be tested compared to a waiting group. Primary outcome variable is the difference in glycemic control between baseline and the 6-month follow-up. Secondary outcome variables are: time-in-range, frequency and duration of hypo- and hyperglycemic episodes, diabetes-related distress, depressive symptoms, health-related quality of life, diabetes self-efficacy, self-care behavior, and hypoglycemia awareness.

DETAILED DESCRIPTION:
The investigators developed a new psychoeducational treatment and education program - called FLASH - for diabetic patients on an intensive insulin therapy who use flash glucose monitoring (FGM).

FLASH is a self-management-based treatment and education program. It is designed to empower patients to adequately use FGM in daily life and to train patients how to analyze their glucose data. FLASH consists of four lessons (90 minutes each).

FLASH is tested in a randomized controlled trial (RCT) with a waiting-list control group since no certified and effective treatment and education program for FGM exists.

This study is a multi-center study. Study centers are specialized diabetes practices throughout Germany. Patients will be approached by their respective practice and informed about the study. Study measurements as well as the conduct of FLASH will take place at the respective practice.

Baseline measurement will take place prior to the beginning of FLASH. After completion of baseline measurement, all patients from one study center will be randomized centrally by the Research Institute of the Diabetes Academy Mergentheim (FIDAM). 2 weeks and 6 months after the completion of FLASH, follow-up measurements will be conducted at the respective study center.

HbA1c as a marker of glycemic control will be analyzed in a central laboratory. Time-in-range and the frequency and duration of hypo- and hyperglycemic episodes will be assessed via stored glucose data on patients FGM devices. The other secondary outcome measures will be assessed via psychometrically tested questionnaires or via patient files.

ELIGIBILITY:
Inclusion Criteria:

* Intensified insulin therapy / insulin pump therapy
* previous participation in a structured diabetes education program
* HbA1c ≥ 7,5% but ≤ 14%
* Reduction of HbA1c as therapeutic goal
* Indication for using FGM
* Ability to understand, speak and write German language
* informed consent (if necessary, informed consent of the parents)

Exclusion Criteria:

* Diabetes duration < 1 year
* Type 2 diabetes without insulin or non-intensified insulin therapy
* severe organic disease preventing a regular participation in the training course
* pregnancy
* severe cognitive impairment
* current treatment of psychiatric disorder
* renal disease requiring dialysis

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Changes in Glycemic Control Measured by A1c | 6 months
  Difference between baseline A1c and A1c at the 6-month follow-up

SECONDARY OUTCOMES:
Changes in "time-in-range" | 6 months
  Difference in the duration of glycemic values spent between 70 mg/dl and 180 mg/dl between baseline and the 6-month follow-up
Changes in hypoglycemic episodes | 6 months
  Differences between the frequency of hypoglycemic glucose values (<70 mg/dl) (baseline vs. follow-up)
Changes in the duration of hypoglycemic episodes | 6 months
  Differences between the duration of hypoglycemic glucose values (<70 mg/dl) (baseline vs. follow-up)
Changes in hyperglycemic episodes | 6 months
  Differences between the frequency of hyperglycemic glucose values (>180 mg/dl) (baseline vs. follow-up)
Changes in the duration of hyperglycemic episodes | 6 months
  Differences between the duration of hyperglycemic glucose values (>180 mg/dl) (baseline vs. follow-up)
Hypoglycaemia Awareness | 6 months
  The hypoglycemia awareness questionnaire provides a score indicating the severity of hypoglycaemia unawareness. This scale ranges from 0 (maximum hypoglycaemia awareness) to 7 (minimum hypoglycaemia awareness), where a score of 4 suggests reduced hypoglycaemia awareness.
Diabetes Empowerment | 6 months
  Empowerment is measured by a German version of the Diabetes Empowerment Scale, a measure of diabetes-related psychosocial self-efficacy.
Diabetes Distress | 6 months
  The Diabetes Distress Scale (DDS-28) assesses diabetes-related stressors due to living and treating diabetes. Different aspects of distress are covered such as hypoglycemia-related distress, physician-related distress
Problem Areas in Diabetes | 6 months
  The Problem Areas in Diabetes Scale (PAID) assesses the psychosocial adaptation to the burden of living with and treating diabetes.
Depressive symptoms | 6 months
  The presence and extent of typical depressive symptoms are assessed via self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Hermanns, PhD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim (FIDAM GmbH)
Locations (1):
- Diabetes und Stoffwechselpraxis Wetter, Wetter, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hermanns N, Ehrmann D, Schipfer M, Kroger J, Haak T, Kulzer B. The impact of a structured education and treatment programme (FLASH) for people with diabetes using a flash sensor-based glucose monitoring system: Results of a randomized controlled trial. Diabetes Res Clin Pract. 2019 Apr;150:111-121. doi: 10.1016/j.diabres.2019.03.003. Epub 2019 Mar 4. PMID 30844467
- [Derived] Schipfer M, Albrecht C, Ehrmann D, Haak T, Kulzer B, Hermanns N. Makes FLASH the difference between the intervention group and the treatment-as-usual group in an evaluation study of a structured education and treatment programme for flash glucose monitoring devices in people with diabetes on intensive insulin therapy: study protocol for a randomised controlled trial. Trials. 2018 Feb 5;19(1):91. doi: 10.1186/s13063-018-2479-9. PMID 29402319